CLINICAL TRIAL: NCT04696419
Title: Measuring the Effects of Different Intensities of Contact to Dogs
Brief Title: Measuring Effects of Contact to Dogs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ANIMAL CONTACT1; 128534 (Other Grant/Funding Number: TrygFonden)
Record Dates: First submitted 2020-10-09; First posted 2021-01-06 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2020-10

CONDITIONS: Physiological Responses to Contact With Dogs; Psychological Responses to Contact With Dogs; Behavioural Responses to Contact With Dogs
Keywords: Animal-assisted therapy; Non-invasive measure; Human-animal contact

STUDY DESIGN:
Intervention Model Description: Randomised within-subject design. Each subject is exposed to three different levels of contact with a dog and a control situation in randomised order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ANIMAL CONTACT 1 (Other): Only one arm - within-subject design
  Interventions: Other: Different intensities of contact to dogs

INTERVENTIONS:
Other: Different intensities of contact to dogs — Each subject is exposed to four test situations of 10 minutes. Three situations with increasing intensity of dog contact, and one control test situation with no contact to a dog. The order of the test situations is random and with 30 minute washout in-between

SUMMARY:
The study aims to identify and quantify objective non-invasive measures of the immediate effect of contact with dogs in a standardized experimental setup. Employing a within-subject design, the study includes healthy participants that are exposed to three different levels of contact to a dog compared with a no-dog control condition while obtaining measures of both physiological, behavioral, and psychological effects.

DETAILED DESCRIPTION:
Using a within-subjects design, we will compare four standardised and controlled test situations with different levels of dog contact:

1) visual (V), 2) tactile and visual (TV), 3) tactile, visual, interaction (TVI), and 4)control (C).

The participants will be subjected to all four test situations on the same day, and will be randomly allocated to test order.

On the test day, we collect background information and baseline measures for the participants (baseline period, duration: 50 minutes), whereafter they rest for 30 minutes (pre-intervention rest period). After this the participants are subjected to the four test situations (10 minutes each) that are followed by rest intervals (30 minutes each).

The participants' interaction with the dog during the 10-minute test situations are standardised according to the specific contact treatment. Most physiological and all behavioural measures are recorded continuously throughout each test in order for us to link the "dosage" of dog (the different levels of contact) with the psychological responses and some physiological measures obtained before an after each test situation.

Below is shown the exact time schedule of the test day, that we refer to when describing the outcome measures. The baseline period (30 minutes) is not included in the total test period (total duration= 190 minutes), that consist of a pre-intervention and intervention period.

* Baseline period (50 minutes - not part of total test period)
* Pre-intervention period (start, t=0 minutes; end t= 30 minutes)
* Test situation 1 (start, t=30 minutes; end, t=40 minutes)
* Rest period 1 (start, t=40 minutes, end, t= 70 minutes)
* Test situation 2 (start, t=70 minutes; end, t=80 minutes)
* Rest period 2 (start, t=80 minutes, end, t= 110 minutes)
* Test situation 3 (start, t=110 minutes; end, t=120 minutes)
* Rest period 3 (start, t=120 minutes, end, t= 150 minutes)
* Test situation 4 (start, t=150 minutes; end, t=160 minutes)
* Rest period 4 (start, t=160 minutes, end, t= 190 minutes)

ELIGIBILITY:
Inclusion Criteria:

* Normal cognitive functioning and physical movement
* Ability to speak and read Danish

Exclusion Criteria:

* Known medical, psychiatric or neurological disease
* Use of psychotropic medications
* Frequent use of pain medication
* Use of illegal psychotropic drugs
* Known allergies to dogs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Physiological measure, heart rate | Measured continuously throughout the total test period of 190 minutes (through the pre-intervention period, the four test situations and all resting periods)
  The test person wears self-adhesive electrodes and the heart rate is measured non-invasively,
Physiological measure, blood pressure | Baseline: Measured at onset of the 30 minute pre-intervention period preceeding the first of the four test situations (t=0 minutes)
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Physiological measure, blood pressure | Test periods: Measured immediately preceeding the first test situation: t=30 minutes
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Physiological measure, blood pressure | Test periods: Measured immediately following the first test situation: t= 40 minutes
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Physiological measure, blood pressure | Test periods: Measured immediately preceeding the second test situation: t= 70 minutes
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Physiological measure, blood pressure | Test periods: Measured immediately following the second test situation: t= 80 minutes
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Physiological measure, blood pressure | Test periods: Measured immediately preceeding the third test situation: t= 110 minutes.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Physiological measure, blood pressure | Test periods: Measured immediately following the third test situation: t= 120 minutes.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Physiological measure, blood pressure | Test periods: Measured immediately preceeding the fourth test situation: t= 150 minutes.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Physiological measure, blood pressure | Test periods: Measured immediately following the fourth test situation: t=160 minutes.
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Physiological measure, blood pressure | After the last resting period: Measured at the end of the last resting period, following the last of the four test situations: t= 190 minutes
  Blood pressure is measured manually with a blood pressure monitor with a blood pressure cuff
Physiological measure, heart rate variablility | Measured continuously throughout the total test period of 190 minutes (through the pre-intervention period, the four test situations and all resting periods)
  Heart rate variability is calculated from heart rate data
Physiological measure, galvanic skin response | Measured continuously throughout the total test period of 190 minutes (through the pre-intervention period, the four test situations and all resting periods)
  The test person is fitted with electrodes on two fingers and galvanic skin response is measured non-invasively,
Salivary cortisol | Baseline: Measured at onset of the 30 minute pre-intervention period preceeding the first of the four test situations (t=0 minutes)
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary cortisol | Test periods: Measured immediately preceeding the first test situation: t=30 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary cortisol | Test periods: Measured immediately following the first test situation: t=40 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary cortisol | Test periods: Measured immediately preceeding the second test situation: t=70 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary cortisol | Test periods: Measured immediately following the second test situation: t=80 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary cortisol | Test periods: Measured immediately preceeding the third test situation: t=110 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary cortisol | Test periods: Measured immediately following the third test situation: t=120 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary cortisol | Test periods: Measured immediately preceeding the fourth test situation: t=150 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary cortisol | Test periods: Measured immediately following the fourth test situation: t=160 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary cortisol | After the last resting period: Measured at the end of the last resting period, following the last of the four test situations; t= 190 minutes
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary oxytocin | Baseline: Measured at onset of the 30 minute pre-intervention period preceeding the first of the four test situations (t=0 minutes)
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary oxytocin | Test periods: Measured immediately preceeding the first test situation: t=30 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary oxytocin | Test periods: Measured immediately following the first test situation: t= 40 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary oxytocin | Test periods: Measured immediately preceeding the second test situation: t= 70 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary oxytocin | Test periods: Measured immediately following the second test situation: t= 80 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary oxytocin | Test periods: Measured immediately preceeding the third test situation: t= 110 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary oxytocin | Test periods: Measured immediately following the third test situation: t= 120 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary oxytocin | Test periods: Measured immediately preceeding the fourth test situation: 150 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary oxytocin | Test periods: Measured immediately following the fourth test situation: t=160 minutes.
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Salivary oxytocin | After the last resting period: Measured at the end of the last resting period, following the last of the four test situations; t= 190 minutes
  Saliva is obtained from the testperson with a cotton swab which is chewed for one minute
Visual analogue scales measuring expected psychological and physiological effects of the test day including, including all four test situations | Baseline: Measured at onset of the 30 minute pre-intervention period preceeding the first of the four test situations (t=0 minutes)
  Test persons fill in a visual analoque scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring expected psychological and physiological effects of each of the four test situations | Test periods: Measured immediately preceeding the first test situation: t=30 minutes
  Test persons fill in a visual analoque scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring expected psychological and physiological effects of each of the four test situations | Test periods: Measured immediately preceeding the second test situation: t= 70minutes
  Test persons fill in a visual analoque scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring expected psychological and physiological effects of each of the four test situations | Test periods: Measured immediately preceeding the third test situation: t= 110 minutes
  Test persons fill in a visual analoque scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring expected psychological and physiological effects of each of the four test situations | Test periods: Measured immediately preceeding the fourth test situation: t=150 minutes
  Test persons fill in a visual analoque scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring perceived psychological and physiological effects of each of the four test situations | Test periods: Measured immediately following the first test situations: t=40 minutes
  Test persons fill in a visual analoque scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring perceived psychological and physiological effects of each of the four test situations | Test periods: Measured immediately following the second test situation: t= 80 minutes
  Test persons fill in a visual analoque scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring perceived psychological and physiological effects of each of the four test situations | Test periods: Measured immediately following the third test situation: t=120 minutes
  Test persons fill in a visual analoque scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring perceived psychological and physiological effects of each of the four test situations | Test periods: Measured immediately following the fourth test situation: t= 160 minutes
  Test persons fill in a visual analoque scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
Visual analogue scales measuring perceived psychological and physiological effects of of the test day including, including all four test situations | After last resting period: Measured at the end of the last resting period, following the last of the four test situations, t=190 minutes
  Test persons fill in a visual analoque scale. Minimum value -100 (very negative effect) and maximum value 100 (very positive effect), and 0 being neutral.
The State-Trait Anxiety Inventory (STAI) | Baseline: Measured at onset of the 30 minute pre-intervention period preceeding the first of the four test situations (t=0 minutes)
  State anxiety is measured with the STAI-scale (minimum score= 20, maximum score= 80, and a lower score indicates a high anxiety level)
The State-Trait Anxiety Inventory (STAI) | Test periods: Measured immediately following the first test situation: t=40 minutes
  State anxiety is measured with the STAI-scale (minimum score= 20, maximum score= 80, and a lower score indicates a high anxiety level)
The State-Trait Anxiety Inventory (STAI) | Test periods: Measured immediately following the second test situation: t= 80 minutes
  State anxiety is measured with the STAI-scale (minimum score= 20, maximum score= 80, and a lower score indicates a high anxiety level)
The State-Trait Anxiety Inventory (STAI) | Test periods: Measured immediately following the third test situation: t= 120 minutes
  State anxiety is measured with the STAI-scale (minimum score= 20, maximum score= 80, and a lower score indicates a high anxiety level)
The State-Trait Anxiety Inventory (STAI) | Test periods: Measured immediately following the fourth test situation: t= 160 minutes
  State anxiety is measured with the STAI-scale (minimum score= 20, maximum score= 80, and a lower score indicates a high anxiety level)
The Positive and Negative Affect Schedule (PANAS) | Baseline: Measured at onset of the 30 minute pre-intervention period preceeding the first of the four test situations (t=0 minutes)
  Positive and negative affect is measured with the PANAS scale, where the person scores whether or not they experience each of 20 emotions on a 5-step scale from "very little /not at all" to "extremely much". The emotions differ in valens.
The Positive and Negative Affect Schedule (PANAS) | Test periods: Measured immediately following the first test situation: t= 40 minutes
  Positive and negative affect is measured with the PANAS scale, where the person scores whether or not they experience each of 20 emotions on a 5-step scale from "very little /not at all" to "extremely much". The emotions differ in valens.
The Positive and Negative Affect Schedule (PANAS) | Test periods: Measured immediately following the second test situation: t= 80 minutes
  Positive and negative affect is measured with the PANAS scale, where the person scores whether or not they experience each of 20 emotions on a 5-step scale from "very little /not at all" to "extremely much". The emotions differ in valens.
The Positive and Negative Affect Schedule (PANAS) | Test periods: Measured immediately following the third test situation: t=120 minutes
  Positive and negative affect is measured with the PANAS scale, where the person scores whether or not they experience each of 20 emotions on a 5-step scale from "very little /not at all" to "extremely much". The emotions differ in valens.
The Positive and Negative Affect Schedule (PANAS) | Test periods: Measured immediately following the fourth test situation: t=160 minutes
  Positive and negative affect is measured with the PANAS scale, where the person scores whether or not they experience each of 20 emotions on a 5-step scale from "very little /not at all" to "extremely much". The emotions differ in valens.

SECONDARY OUTCOMES:
Quantitative behavioural measures - frequencies of behavioural elements | Measured continuously throughout the total test period of 190 minutes (through the pre-intervention period, the four test situations and all resting periods)
  A video recording of the test persons behaviour is analysed for frequency of predefined behavioural elements Postures: sitting, standing walkning Touching the dog: being in physical contact with the dog with tha hand or another part of the body Looking at the dog: Having head turned towards the dog Talking to the dog: Directing talk directly at the dog, as opposed to the person present
Quantitative behavioural measures - duration of behavioural elements | Measured continuously throughout the total test period of 190 minutes (through the pre-intervention period, the four test situations and all resting periods)
  A video recording of the test persons behaviour is analysed for the duration (seconds) of predefined behavioural elements Postures: sitting, standing walkning Touching the dog: being in physical contact with the dog with tha hand or another part of the body Looking at the dog: Having head turned towards the dog Talking to the dog: Directing talk directly at the dog, as opposed to the person present

CONTACTS AND LOCATIONS:
Overall Officials: Karen Thodberg, Principal Investigator — Senior researcher
Locations (1):
- Aarhus University, Tjele, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fuglsang-Damgaard LH, Lunde SJ, Christensen JW, Vase L, Videbech PB, Thodberg K. Human physiological responses to different types of human-dog interactions: A randomised crossover study. Complement Ther Clin Pract. 2024 Nov;57:101899. doi: 10.1016/j.ctcp.2024.101899. Epub 2024 Aug 26. PMID 39217835